CLINICAL TRIAL: NCT02519439
Title: A follow-on, Two-year Open-label Extension Study of Ganaxolone as add-on Therapy in Adult Patients With Drug-resistant Partial-onset Seizures
Brief Title: A Two-year Open-label Extension Study of Ganaxolone in Patients With Drug-resistant Partial-onset Seizures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Ganaxolone missed its primary endpoint in the double-blind portion of the 1042-0603 study. Due to this outcome Marinus discontinued this extension study.
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1042-0604
Record Dates: First submitted 2015-06-04; First posted 2015-08-11 (Estimated); Results first posted 2023-02-14 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Drug Resistant Partial Onset Seizure
Keywords: Partial Onset Seizures; complex partial seizures; simple partial seizures; anticonvulsant; ganaxolone; neurosteroid; Marinus; epilepsy
MeSH Terms: conditions — Seizures; Epilepsies, Partial; Epilepsy | interventions — ganaxolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ganaxolone (Experimental): Up to a maximum of 1800 mg/day
  Interventions: Drug: ganaxolone

INTERVENTIONS:
Drug: ganaxolone — 225 mg capsules 450 mg to 900 mg 2x/day
  Other Names: CCD 1042

SUMMARY:
A follow-on, two-year open-label extension study of ganaxolone as add-on therapy in adult patients with drug-resistant partial-onset seizures

DETAILED DESCRIPTION:
This study is a 2-year, open-label continuation for those patients benefiting from ganaxolone treatment after completing Protocol 1042-0603.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed all scheduled clinical study visits in the previous protocol 1042-0603 and have shown a minimum 35% improvement in mean 28-day seizure frequency over the last three 28-day periods in study 1042-603 as compared to the baseline of study 1042-603.
* Subjects whose daily study drug compliance in Study 1042-0603 was 90% or greater, and for whom the investigator feels that the subject was compliant with the full dose as prescribed.
* Able to give informed consent in writing, or have a legally authorized representative able to do so, after being properly informed of the nature and risks of the study and prior to engaging in any study-related procedures.
* Currently being treated and maintained with a stable regimen of 1, 2, or 3 anti-epileptic drugs (AED) at a consistent dose for one month prior to study entry.
* Implanted Vagus Nerve Stimulator (VNS) is permitted and will not count towards the number of concomitant AEDs.
* Able and willing to maintain an accurate and complete daily written seizure calendar or has a caregiver who is able and willing to maintain an accurate and complete daily written seizure calendar.
* Able and willing to take drug with food twice daily. Ganaxolone must be administered with food.
* Sexually active women of childbearing potential (WCBP) must be using a medically acceptable method of birth control and have a negative pregnancy test at Visit 1 and at subsequent visits.

Exclusion Criteria:

* Have any medical condition that, in the investigator's judgment, is considered to be clinically significant and could potentially affect subject safety or study outcome
* Experienced a Serious Adverse Event or a moderate or severe medically important adverse event judged probably or definitely related to open-label ganaxolone in the previous study, 1042-0603
* Have Alanine transferase (ALT; SGPT) or Aspartate transferase (AST; SGOT) levels > 3 times upper limits of normal (ULN), or total bilirubin >1.5 time ULN during Study 1042-0603.
* Have a history of malignancy within the past 2 years, with the exception of basal cell carcinoma.
* Seizures secondary to illicit drug or alcohol use, infection, neoplasm, demyelinating disease, degenerative neurological disease, or central nervous system (CNS) disease deemed progressive, metabolic illness, or progressive degenerative disease.
* Have active suicidal plan/intent, or have had active suicidal thoughts in the past 6 months. Have a history of an actual suicide attempt in the last 5 years or more than 1 lifetime actual suicide attempt as classified by the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Have a history of drug or alcohol abuse within the past 5 years. As with other AEDs, the use of alcohol is not advised.
* Are currently following or planning to follow a ketogenic diet.
* Current use of vigabatrin or ezogabine (retigabine; Potiga; Trobalt) is not permitted.
* Females who are pregnant, currently breastfeeding or planning to become pregnant during the study.
* Inability/unwillingness to withhold grapefruit and grapefruit juice from diet during the entire clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Neurological Research Institute, Santa Monica, California
  - Bluegrass Epilepsy Research, LLC, Lexington, Kentucky
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Texas Epilepsy Group, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label extension of Study 1042-0603, providing a two-year adjunctive ganaxolone treatment to adult participants with epilepsy consisting of partial-onset seizures (POS).
Pre-assignment Details: A total of 26 participants moved in from 1042-0603 (NCT01963208) study. As Ganaxolone missed its primary endpoint in the double-blind portion of the 1042-0603 study, the study was terminated.
Groups:
- Ganaxolone: Participants entered the study at their current dose of ganaxolone (450 milligrams [mg] to 900 mg twice daily; up to a maximum dose of 1800 mg per day) from Study 1042-0603 (NCT01963208). The dose of ganaxolone has been adjusted for tolerability and response.
Period: Overall Study
Arm/Group | Ganaxolone
Started | 26
Completed | 5
Not Completed | 21
Not completed — Study Termination | 19
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who signed informed consent and took one dose of study medication in this study.
Arm/Group | Ganaxolone
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.3 (15.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in 28-day Seizure Frequency
Description: Baseline 28-day seizure frequency was calculated as the number of seizures in the Baseline period of Study 1042-0603 (less than or equal to 56 days) divided by the number of days with available seizure data in the Baseline period and multiplied by 28. Post-baseline 28-day seizure frequency was calculated as the number of seizures in the entire treatment period divided by the number of days with available seizure data in the treatment period and multiplied by 28. Baseline was defined as the last non-missing value obtained before the first treatment in the preceding Study 1042-0603. The calculation for percent change from Baseline in 28-day seizure frequency was done as follows for each participant: post-Baseline 28-day seizure frequency minus Baseline 28-day seizure frequency whole divided by Baseline 28-day seizure frequency multiplied by 100 percent.
Time Frame: Baseline and at Day 28
Population: Full Analysis Population included participants who returned at least 25 days of seizure calendar data.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ganaxolone
Number analyzed (Participants) | 26
Percent change | -41.86 (44.913)

2. Secondary Outcome: Number of Participants Who Showed Greater Than or Equal to 50% Reduction in 28-day Seizure Frequent From Baseline
Description: A 50% responder is an individual whose reduction of percent change from Baseline to the end of the open label extension period in 28-day partial-onset seizure (POS) seizure frequency is greater than or equal to 50%.
Time Frame: Baseline and at Day 28
Population: Full Analysis Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone
Number analyzed (Participants) | 26
Participants | 14

3. Secondary Outcome: Number of Participants With Clinical Global Impression of Improvement (CGI-I) Scores
Description: The CGI-I scale is a clinician-rated 7-point scale used to assess how much the participant's illness had improved or worsened relative to a Baseline state at the beginning of the intervention. It was rated as: 1. "very much improved" 2. "much improved" 3. "minimally improved" 4. "no change" 5. "minimally worse" 6. "much worse" 7. "very much worse". Higher scores indicated worse condition. Participants who showed CGI improvement at Week 104 (End of treatment) has been presented.
Time Frame: At Week 104
Population: Safety Population included all participants who signed informed consent and took one dose of study medication in this study. Only those participants with data available at indicated timepoints has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone
Number analyzed (Participants) | 23
Participants
  Very much improved | 1
  Much improved | 9
  Minimally improved | 11
  No change | 2
  Minimally worse | 0
  Much worse | 0
  Very much worse | 0

4. Secondary Outcome: Number of Participants With Patient/Caregiver Global Impression of Improvement (PGI-I) Scores
Description: The participant is asked to rate the total improvement of their partial-onset seizures whether or not in the participant's judgment it is due entirely to drug treatment based on a 7-point scale using the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse, or very much worse" (1 = very much improved; 7 = very much worse). Higher scores indicated worse condition. Participants who showed PGI improvement at Week 104 (End of treatment) has been presented.
Time Frame: At Week 104
Population: Safety Population. Only those participants with data available at indicated time points has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone
Number analyzed (Participants) | 23
Participants
  Very much improved | 4
  Much improved | 8
  Minimally improved | 10
  No change | 1
  Minimally worse | 0
  Much worse | 0
  Very much worse | 0

ADVERSE EVENTS:
Time Frame: Up to Week 104
Description: Adverse events and Serious adverse events were collected in Safety Population.
Arm/Group | Ganaxolone
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 10/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=26)
Pulmonary embolism/ (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=26)
Headache (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Cellulitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Lip injury (Injury, poisoning and procedural complications) | 1
Lacrimal disorder (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Hepatic enzyme increased (Investigations) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Insomnia (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT02519439/Prot_002.pdf
  • Statistical Analysis Plan (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT02519439/SAP_001.pdf